CLINICAL TRIAL: NCT04658277
Title: Effect of Long Term Clarithromycin for Prevention of Exacerbations in Non-cystic Fibrosis Bronchiectasis in Asian Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Macrolid/Bronchiectasis/2019
Record Dates: First submitted 2020-08-31; First posted 2020-12-08 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Bronchiectasis Adult
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Patients will be given one tab of Clarithromycin 250mg daily.
  Interventions: Drug: Clarithromycin
- usual care (Placebo Comparator): Patients will receive usual medical care
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Clarithromycin — Patients in the intervention arm will take Clarithromycin 250mg daily.
  Arms: Treatment
Other: Usual care — Patients will receive usual medical care
  Arms: usual care

SUMMARY:
clarithromycin may reduce the exacerbations in middle-aged and elderly patients with non-CF bronchiectasis.

The study is aimed to (A) investigate the etiologies and clinical features of patients with bronchiectasis, (B) compare the effect of clarithromycin 250mg daily on the frequency of exacerbations, quality of life and lung function, stratified according to the degree of bronchiectasis severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 years or older
* At least 2 or more exacerbation requiring antibiotic treatment in the past year Clinically stable for at least 4 weeks prior to enrollment (defined as no symptoms of exacerbation, no requirement for supplemental antibiotic therapy)
* Diagnosis of bronchiectasis defined by high-resolution computed tomography (CT) scan

Exclusion Criteria:

* History of cystic fibrosis; hypogammaglobulinemia; allergic bronchopulmonary aspergilosis,
* Cigarette smoking within 6 months
* A positive culture of non-tuberculosis mycobacteria in the past 2 years or at screening
* Macrolide treatment for more than 3 months in the past 6 months
* Oral or intravenous courses of corticosteroids within 30 days of screening
* Any antimicrobial treatment for lower respiratory tract infection in the last 2 weeks
* Unstable arrhythmia
* History of coronary artery disease, or symptoms of heart disease
* Known allergy or intolerance to macrolides
* Patients with liver disease or with elevated transaminanse (aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels equal to or greater than the upper limit of the normal)
* Concurrent medication: Colchicine, calcium channel blocker, statins, amiodarone, amitriptyline, trazodone, citalopram, disopyramide, itraconazole, saquinavir, ritaonavir, atazanavir, sildenafil, tadalafil, vardenafil, theophylline, carbamazepine.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
number of infectious exacerbations | 26 weeks

SECONDARY OUTCOMES:
Time to first exacerbation (Days) | 26 weeks
Rate of symptom-based exacerbations (number of events per month) | 26 weeks
change of post bronchodilator Forced Expiratory volume in 1 sec and forced vital capacity | 26 weeks
change of exercise capacity (flights of stairs) | 26 weeks
change of St George Respiratory Questionnaire Score | 26 weeks
  Scores range from 0 to 100, with higher scores indicating more limitations.
change of concentration of serum c-reactive protein (mg/L) | 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong, Hong Kong, Please Select, Hong Kong

IPD SHARING:
Plan to Share IPD: No